CLINICAL TRIAL: NCT02276508
Title: Phase 1 Open Label Trial of Nissle 1917 to Assess Safety and Tolerance in Healthy Adult Volunteers
Brief Title: Open Label Trial of Nissle 1917
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elizabeth Lucas (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Lucas, Principal Invesgator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IRB14-00586
Record Dates: First submitted 2014-10-23; First posted 2014-10-28 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotic (Experimental): Participants will take the E. coli Nissle 1917 as an orally administered medication first while in clinic to be observed for 30 minutes for any hypersensitivity reaction. The dose of Nissle 1917 will be 100mg capsule (2.5-25x109 organism) once daily for a total of 4 days. Participants will then increase the dose to 2 capsules (200mg) once daily for the remaining 26 days of the study period.
  Interventions: Drug: E. coli Nissle 1917

INTERVENTIONS:
Drug: E. coli Nissle 1917 — Participants will all take E. coli Nissle 1917 orally administered medication for 30 days
  Other Names: Mutaflor

SUMMARY:
Nissle 1917 is an E. coli based probiotic used in the Europe for close to 100 years to treat gastrointestinal disorders and infections. The investigators will assess the safety and tolerability of this medication in Americans in a Phase 1 trial.

DETAILED DESCRIPTION:
Background: Nissle 1917 is an E. coli based probiotic that has been successfully used in Europe for close to 100 years to treat largely gastrointestinal disorders like inflammatory bowel disease, gastroenteritis, and irritable bowel syndrome. In addition to those disorders, we believe that Nissle 1917 is a promising alternative therapy for prevention of urinary tract infections in susceptible individuals.

Purpose: The Phase 1 trial will use Nissle 1917 in healthy adult patient volunteers for the first time in the United States. The investigators will track the frequency and incidence of side effects and adverse events.

Participants:

20 adult (>21 years of age) healthy volunteers

Protocol:

* Participants will enroll in our trial after a review of medical history and physical.
* Participants will then take 30 day course of Nissle 1917 capsules
* Investigators will telephone participants 1-2 weeks after they have begun the trial to assess for any side effects or adverse events
* Subjects will also be provided with a diary to record any side effects or adverse events
* At the end of 30 days, participants will return to clinic for a follow up visit to discuss any side effects or adverse events experienced during the trial and to return any unused medication
* Investigators will again telephone all participants 28-35 days following completion of the study drug again to pose a questionnaire aimed at revealing any side effects or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer of age 21 years or older

Exclusion Criteria:

* Any individual with an active urinary tract infection (UTI)
* Any individual with an acute illness within the past 7 days
* Any individual with neurogenic bladder or with vesicoureteral reflux
* Any individual with any anatomic abnormality, congenital or acquired, of the urinary tract system
* Any individual with any anatomic abnormality, congenital or acquired, of the gastrointestinal tract
* Any individual with untreated dysfunctional elimination syndrome
* Immunocompromised patients
* Individuals with a central venous catheter
* Individuals requiring the use of antibiotics, immunomodulatory medications, or other probiotics
* Any participant with a history of chronic gastrointestinal disease
* Any individual with a chronic uncontrolled medical illness
* Any female of reproductive age who is currently pregnant, breastfeeding, or sexually active and unwilling or unable to use an acceptable method of contraception.
* Any participant is unable to appropriately take and store medication
* Any individual enrolled in a clinical trial evaluating another investigational agent in the last 30 days.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events associated with ingestion of E. coli Nissle 1917 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Venkata R Jayanthi, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States